CLINICAL TRIAL: NCT07017465
Title: Determination of the Glycemic Index (GI) and Glycemic Load (GL) of Watermelon (Citrullus Lanatus) in Healthy Adults (A Controlled Clinical Trial)
Brief Title: Determination of the Glycemic Index (GI) and Glycemic Load (GL) of Watermelon (Citrullus Lanatus) in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Naseer Ahmed, Associate Professor, Rehman Medical Institute - RMI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GL/GI-NA_1V3
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Glycemic Index; Glycemic Load
Keywords: GLYCEMIC INDEX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (cross over) (Active Comparator): Participants will consume a standard oral glucose solution containing 50 grams of available carbohydrate. This serves as the reference for calculating glycemic index.
  Interventions: Other: Water melon (sugar baby); Other: watermelon (Charleston gray); Other: watermelon (Crimson sweet)

INTERVENTIONS:
Other: Water melon (sugar baby) — Participants will consume a portion of watermelon Type A containing 50 grams of available carbohydrate to evaluate its glycemic index and glycemic load.
Other: watermelon (Charleston gray) — Participants will consume a portion of watermelon Type B containing 50 grams of available carbohydrate to evaluate its glycemic index and glycemic load.
Other: watermelon (Crimson sweet) — Participants will consume a portion of watermelon Type C containing 50 grams of available carbohydrate to evaluate its glycemic index and glycemic load.

SUMMARY:
This study aims to evaluate and compare the glycemic load (GL) and glycemic index (GI) of different types of watermelons commonly available in the market. Using glucose as the reference standard, the study will measure the blood glucose response following consumption of each watermelon type in healthy adult participants.

DETAILED DESCRIPTION:
his study aims to evaluate and compare the glycemic load (GL) and glycemic index (GI) of different types of watermelons commonly available in the market. Using glucose as the reference standard, the study will measure the blood glucose response following consumption of each watermelon type in healthy adult participants. The objective is to identify variations in glycemic impact among watermelon varieties to inform dietary recommendations for blood sugar management.

ELIGIBILITY:
Inclusion Criteria:•

1. Healthy adults (BMI 18.5-24.9kg/m2.
2. No history of diabetes or metabolic disorders.
3. Not taking any medication affecting glucose metabolism.

Exclusion Criteria:

1) GI Disorders. 2) Recent infections or illness affecting glucose tolerance. 3) Non willing participants.

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index (GI) of Watermelon Varieties | 1 month
  Description: Incremental area under the blood glucose response curve (iAUC) over 120 minutes after consuming each watermelon type, expressed as a percentage of the iAUC after consuming the glucose reference.

SECONDARY OUTCOMES:
Glycemic Load (GL) of Watermelon Varieties | 1 month
  Calculated using the formula:
  Glycemic Load = (GI × carbohydrate content per typical serving) ÷ 100

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] A. Coughlan , E. Anderson , L. Stern , A. El-Ansary , in: Marketing Channels, Prentice Hall, New Jersey, 2001, p. 590p .
- [Background] R. Clodius , W. Mueller , Market structure analysis, an orientation for research in agricultural economics, J. Farm Econ. 43 (3) (1961) 513-553 .
- [Background] A. Camelo , in: Manuel Pour La Préparation Et La Vente Des Fruits Et Des Légumes Du Champ Au Marché, Bulletin des Services Agricoles de la FAO. FAO, Rome, 2007, p. 205 p .
- [Background] I. Adeoye , T. Olajide , A. Adebisi , J. Usman , M. Badmus , Economic analysis of watermel on based production system in Oyo state, J. Agric. Biol. Sci. 6 (7) (2011) 53-59 .
- [Background] E.G. Achigan-Dako , R. Fagbemissi , H.T. Avohou , R.S. Vodouhe , O. Coulibaly , A. Ahanchede , Importance and practices of Egusi crops (Citrullus lanatus (Thunb.) Matsum. & Nakai, Cucumeropsis mannii Naudin and Lagenaria siceraria (Molina) Standl. cv. ' Aklamkpa ') in sociolinguistic areas in Benin, Biotechnol. Agron. Soc. Environ. 12 (4) (2008) 393-403 .
- [Background] I.A. Abdou , Modiﬁed marketing eﬃciency criteria for consideration in cropping structure planning: a case of newly reclaimed land farmers in Egypt, in: S. O'reilly, M. Keane, P. Enright (Eds.), Proceedings of the 16th international farm management association congress, a vibrant rural economy-the challenge for balance, Cork Ireland, 2007, pp. 79-84